CLINICAL TRIAL: NCT02440802
Title: Evaluation and Predictive Value of Genetic Polymorphisms in the Management of Hormonal Treatment of Prostate Cancer
Acronym: Feel+
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: B403201317385
Record Dates: First submitted 2015-04-30; First posted 2015-05-12 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — One saliva sample (2mL) will be collected once at baseline for single nucleotide polymorphism analyses.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Gonadoliberin antagonist treatment: Single arm study, all patients are treated the same way. Saliva sample collection for genetic analyses.
  Interventions: Genetic: Saliva sample collection for genetic analyses

INTERVENTIONS:
Genetic: Saliva sample collection for genetic analyses — Patients with Prostate cancer receiving androgen deprivation treatment with a GnRH antagonist will be followed-up for 6 months for quality of life. At Baseline, 3 months and 6 months of treatment QoL data will be collected, as well as body parameters. At Baseline, once, a saliva sample will be collected for genetic analyses.

SUMMARY:
Androgen deprivation therapy (ADT) by surgical castration or administration of LHRH agonists or antagonists is the gold-standard systemic treatment of Prostate Cancer. The efficacy, severity and frequency of side effects of ADT vary from a patient to another. The exact cause of this variability is not known, however certain genetic polymorphisms affecting enzymes implicated in the synthesis and metabolism of sex-steroids seem to be involved in these processes.

To perform a longitudinal study to evaluate the prevalence of various genetic polymorphisms affecting genes in the sex-steroid synthesis and metabolism pathway (CYP1A1, CYP1B1, CYP19A1, 17HSD, HSD3B1, AR, ESR1, ESRRG, IL6, TNF-alpha) in men with Prostate Cancer receiving ADT and the possible association between polymorphisms and frequency and severity of side-effects of ADT.

DETAILED DESCRIPTION:
Prostate cancer patients for which reimbursed ADT with a gonadoliberin antagonist is indicated, for a period of at least 6 months will lbe enrolled. At 0, 3 months and 6 months of ADT, Aging Males' Symptoms (AMS), EQ-5D (EuroQoL), and hot flashes intensity and frequency (Moyad scale) will be collected, as well as routine assessments: vital signs (blood pressure, heart rate), weight, waist perimeter, fat percentage, Body Mass Index (BMI) and routine laboratory assessments. Determine genotypes of polymorphisms of interest by pyrosequencing. Determine the prevalence of the polymorphisms of interest in the studied population. Perform initial assessment of the association between genetic polymorphisms and questionnaire results.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer patients for which reimbursed ADT with a gonadoliberin antagonist is indicated, for a period of at least 6 months.

Exclusion Criteria:

* Prostate cancer patients who are already receiving ADT with a gonadoliberin antagonist.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prostate cancer patients for which reimbursed androgen deprivation therapy with a gonadoliberin antagonist is indicated, for aperiod of at least 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2013-04; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Aging Males Symptoms questionnaire | 0 months
Aging Males Symptoms questionnaire | 3 months
Aging Males Symptoms questionnaire | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand TOMBAL, MD, PhD, Principal Investigator — Cliniques Universitaires Saint Luc, Brussels
Locations (20):
- Belgium (20):
  - ASZ Aalst, Aalst
  - OLV Aalst, Aalst
  - ZNA Middelheim, Antwerp
  - CHu Saint Pierre, Brussels
  - Hopital Erasme, Brussels
  - Cliniques Universitaires Saint Luc, Brussels
  - AZ Sint Blasius, Dendermonde
  - JESSA Ziekenhuis, Hasselt
  - Jan Ypermanziekenhuis, Ieper
  - CHU Tivoli, La Louvière
  - CHR Citadelle, Liège
  - AZ Sint Jozef, Malle
  - ZNA Jan Palfijn, Merksem
  - CH Mouscron, Mouscron
  - Clinique Saint Luc Bouge, Namur
  - AZ Damiaan, Ostend
  - AZ Delta, Roeselare
  - AZ St Jozef, Turnhout
  - AZ Jan Portaels, Vilvoorde
  - CHU Mont-Godinne, Yvoir

REFERENCES:
- [Background] Mottet N, Bellmunt J, Bolla M, Joniau S, Mason M, Matveev V, Schmid HP, Van der Kwast T, Wiegel T, Zattoni F, Heidenreich A. EAU guidelines on prostate cancer. Part II: Treatment of advanced, relapsing, and castration-resistant prostate cancer. Eur Urol. 2011 Apr;59(4):572-83. doi: 10.1016/j.eururo.2011.01.025. Epub 2011 Jan 25. PMID 21315502
- [Background] Mohile SG, Mustian K, Bylow K, Hall W, Dale W. Management of complications of androgen deprivation therapy in the older man. Crit Rev Oncol Hematol. 2009 Jun;70(3):235-55. doi: 10.1016/j.critrevonc.2008.09.004. Epub 2008 Oct 25. PMID 18952456
- [Background] Allain TJ. Prostate cancer, osteoporosis and fracture risk. Gerontology. 2006;52(2):107-10. doi: 10.1159/000090956. PMID 16508318
- [Background] Benton MJ, White A. Osteoporosis: recommendations for resistance exercise and supplementation with calcium and vitamin D to promote bone health. J Community Health Nurs. 2006 Winter;23(4):201-11. doi: 10.1207/s15327655jchn2304_1. PMID 17064230
- [Background] Diamond TH, Higano CS, Smith MR, Guise TA, Singer FR. Osteoporosis in men with prostate carcinoma receiving androgen-deprivation therapy: recommendations for diagnosis and therapies. Cancer. 2004 Mar 1;100(5):892-9. doi: 10.1002/cncr.20056. PMID 14983482
- [Background] McGrath SA, Diamond T. Osteoporosis as a complication of orchiectomy in 2 elderly men with prostatic cancer. J Urol. 1995 Aug;154(2 Pt 1):535-6. doi: 10.1097/00005392-199508000-00057. No abstract available. PMID 7609129
- [Background] Oefelein MG, Ricchuiti V, Conrad W, Seftel A, Bodner D, Goldman H, Resnick M. Skeletal fracture associated with androgen suppression induced osteoporosis: the clinical incidence and risk factors for patients with prostate cancer. J Urol. 2001 Nov;166(5):1724-8. doi: 10.1016/s0022-5347(05)65661-3. PMID 11586210
- [Background] Braga-Basaria M, Dobs AS, Muller DC, Carducci MA, John M, Egan J, Basaria S. Metabolic syndrome in men with prostate cancer undergoing long-term androgen-deprivation therapy. J Clin Oncol. 2006 Aug 20;24(24):3979-83. doi: 10.1200/JCO.2006.05.9741. PMID 16921050
- [Background] Galvao DA, Spry NA, Taaffe DR, Newton RU, Stanley J, Shannon T, Rowling C, Prince R. Changes in muscle, fat and bone mass after 36 weeks of maximal androgen blockade for prostate cancer. BJU Int. 2008 Jul;102(1):44-7. doi: 10.1111/j.1464-410X.2008.07539.x. Epub 2008 Mar 11. PMID 18336606
- [Background] Galvao DA, Taaffe DR, Spry N, Joseph D, Turner D, Newton RU. Reduced muscle strength and functional performance in men with prostate cancer undergoing androgen suppression: a comprehensive cross-sectional investigation. Prostate Cancer Prostatic Dis. 2009;12(2):198-203. doi: 10.1038/pcan.2008.51. Epub 2008 Oct 14. PMID 18852703
- [Background] Smith MR, Lee H, McGovern F, Fallon MA, Goode M, Zietman AL, Finkelstein JS. Metabolic changes during gonadotropin-releasing hormone agonist therapy for prostate cancer: differences from the classic metabolic syndrome. Cancer. 2008 May 15;112(10):2188-94. doi: 10.1002/cncr.23440. PMID 18348297
- [Background] Smith MR, O'Malley AJ, Keating NL. Gonadotrophin-releasing hormone agonists, diabetes and cardiovascular disease in men with prostate cancer: which metabolic syndrome? BJU Int. 2008 Jun;101(11):1335-6. doi: 10.1111/j.1464-410X.2008.07707.x. No abstract available. PMID 18454791
- [Background] D'Amico AV, Denham JW, Bolla M, Collette L, Lamb DS, Tai KH, Steigler A, Chen MH. Short- vs long-term androgen suppression plus external beam radiation therapy and survival in men of advanced age with node-negative high-risk adenocarcinoma of the prostate. Cancer. 2007 May 15;109(10):2004-10. doi: 10.1002/cncr.22628. PMID 17397033
- [Background] D'Amico AV, Denham JW, Crook J, Chen MH, Goldhaber SZ, Lamb DS, Joseph D, Tai KH, Malone S, Ludgate C, Steigler A, Kantoff PW. Influence of androgen suppression therapy for prostate cancer on the frequency and timing of fatal myocardial infarctions. J Clin Oncol. 2007 Jun 10;25(17):2420-5. doi: 10.1200/JCO.2006.09.3369. PMID 17557956
- [Background] D'Amico AV, Loffredo M, Renshaw AA, Loffredo B, Chen MH. Six-month androgen suppression plus radiation therapy compared with radiation therapy alone for men with prostate cancer and a rapidly increasing pretreatment prostate-specific antigen level. J Clin Oncol. 2006 Sep 1;24(25):4190-5. doi: 10.1200/JCO.2006.06.8239. PMID 16943536
- [Background] Efstathiou JA, Bae K, Shipley WU, Hanks GE, Pilepich MV, Sandler HM, Smith MR. Cardiovascular mortality after androgen deprivation therapy for locally advanced prostate cancer: RTOG 85-31. J Clin Oncol. 2009 Jan 1;27(1):92-9. doi: 10.1200/JCO.2007.12.3752. Epub 2008 Dec 1. PMID 19047297
- [Background] Ross RW, Oh WK, Xie W, Pomerantz M, Nakabayashi M, Sartor O, Taplin ME, Regan MM, Kantoff PW, Freedman M. Inherited variation in the androgen pathway is associated with the efficacy of androgen-deprivation therapy in men with prostate cancer. J Clin Oncol. 2008 Feb 20;26(6):842-7. doi: 10.1200/JCO.2007.13.6804. PMID 18281655
- [Background] Jim HS, Park JY, Permuth-Wey J, Rincon MA, Phillips KM, Small BJ, Jacobsen PB. Genetic predictors of fatigue in prostate cancer patients treated with androgen deprivation therapy: preliminary findings. Brain Behav Immun. 2012 Oct;26(7):1030-6. doi: 10.1016/j.bbi.2012.03.001. Epub 2012 Mar 28. PMID 22475653
- [Background] Shearman AM, Cupples LA, Demissie S, Peter I, Schmid CH, Karas RH, Mendelsohn ME, Housman DE, Levy D. Association between estrogen receptor alpha gene variation and cardiovascular disease. JAMA. 2003 Nov 5;290(17):2263-70. doi: 10.1001/jama.290.17.2263. PMID 14600184
- [Background] Alevizaki M, Cimponeriu AT, Garofallaki M, Sarika HL, Alevizaki CC, Papamichael C, Philippou G, Anastasiou EA, Lekakis JP, Mavrikakis M. The androgen receptor gene CAG polymorphism is associated with the severity of coronary artery disease in men. Clin Endocrinol (Oxf). 2003 Dec;59(6):749-55. doi: 10.1046/j.1365-2265.2003.01917.x. PMID 14974917
- [Background] Fox CS, Yang Q, Cupples LA, Guo CY, Atwood LD, Murabito JM, Levy D, Mendelsohn ME, Housman DE, Shearman AM. Sex-specific association between estrogen receptor-alpha gene variation and measures of adiposity: the Framingham Heart Study. J Clin Endocrinol Metab. 2005 Nov;90(11):6257-62. doi: 10.1210/jc.2005-0670. Epub 2005 Sep 6. PMID 16144952
- [Background] Elfassihi L, Giroux S, Bureau A, Laflamme N, Cole DE, Rousseau F. Association with replication between estrogen-related receptor gamma (ESRRgamma) polymorphisms and bone phenotypes in women of European ancestry. J Bone Miner Res. 2010 Apr;25(4):901-11. doi: 10.1359/jbmr.091014. PMID 19821770
- [Background] Crandall CJ, Crawford SL, Gold EB. Vasomotor symptom prevalence is associated with polymorphisms in sex steroid-metabolizing enzymes and receptors. Am J Med. 2006 Sep;119(9 Suppl 1):S52-60. doi: 10.1016/j.amjmed.2006.07.007. PMID 16949389
- [Background] Rodriguez-Gonzalez G, Ramirez-Moreno R, Perez P, Bilbao C, Lopez-Rios L, Diaz-Chico JC, Lara PC, Serra-Majem L, Chirino R, Diaz-Chico BN. The GGN and CAG repeat polymorphisms in the exon-1 of the androgen receptor gene are, respectively, associated with insulin resistance in men and with dyslipidemia in women. J Steroid Biochem Mol Biol. 2009 Feb;113(3-5):202-8. doi: 10.1016/j.jsbmb.2008.12.009. Epub 2008 Dec 30. PMID 19159685
- [Background] Moyad MA. Promoting general health during androgen deprivation therapy (ADT): a rapid 10-step review for your patients. Urol Oncol. 2005 Jan-Feb;23(1):56-64. doi: 10.1016/j.urolonc.2005.03.018. PMID 15885584